CLINICAL TRIAL: NCT06243939
Title: The Effect of Motivational Interviewing on Health Management Self-Efficacy and Quality of Life in Pregnants With Gestational Diabetes Mellitus
Brief Title: The Effect of Motivational Interviewing on Self-Efficacy and Quality of Life in Gestational Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Meltem Akbaş, Assistant Professor, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 02.06.2023/134
Record Dates: First submitted 2023-11-15; First posted 2024-02-06 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Motivational Interviewing; Self Efficacy; Quality of Life; Gestational Diabetes Mellitus
Keywords: Pregnancy; gestational diabetes mellitus; health management self-efficacy; quality of life; motivational interview
MeSH Terms: conditions — Diabetes, Gestational | interventions — Quality of Life

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Education (Experimental): 24-26 weeks for pregnant women diagnosed with gestational diabetes mellitus. A total of motivational interviews will be held for 4 weeks with the pregnant women. Personal Information Form, Health Management Self-Efficacy Scale and Quality of Life Scale will be administered before the motivational interview, and the Health Management Self-Efficacy Scale and Quality of Life Scale will be administered at the end of the motivational interview.
  Interventions: Behavioral: Motivational Interview to Increase Health Management Self-Efficacy and Quality of Life in Pregnant Women Diagnosed with Gestational Diabetes Mellitus
- Control (No Intervention): 24-26 weeks for pregnant women diagnosed with gestational diabetes mellitus. Personal Information Form, Health Management Self-Efficacy Scale and Quality of Life Scale will be applied to the pregnant patient.

INTERVENTIONS:
Behavioral: Motivational Interview to Increase Health Management Self-Efficacy and Quality of Life in Pregnant Women Diagnosed with Gestational Diabetes Mellitus — Motivational interviewing is a client-centered approach used to elicit behavioral change by helping clients explore and resolve their ambivalence.
  Arms: Education

SUMMARY:
This study is a randomized controlled experimental study planned to investigate the effect of motivational interviewing on health management self-efficacy and quality of life in pregnant women with gestational diabetes mellitus.

DETAILED DESCRIPTION:
This study is a randomized controlled experimental study planned to investigate the effect of motivational interviewing on health management self-efficacy and quality of life in pregnant women with gestational diabetes mellitus. 24-26 weeks for pregnant women diagnosed with gestational diabetes mellitus. A total of motivational interviews will be held for 4 weeks with the pregnant women. Personal Information Form, Health Management Self-Efficacy Scale and Quality of Life Scale will be administered before the motivational interview, and the Health Management Self-Efficacy Scale and Quality of Life Scale will be administered at the end of the motivational interview.

ELIGIBILITY:
Inclusion Criteria:

Being pregnant for the first time

* Being diagnosed with gestational diabetes mellitus
* 24-28. Being in the pregnancy week
* Being able to speak and understand Turkish
* Being 18 years or older
* Having a single and viable fetus
* Volunteering to participate in research
* Having and being able to use a mobile phone
* Having all check-ups at the same hospital and regularly throughout pregnancy,

Exclusion Criteria:

* Being diagnosed with diabetes mellitus (type 1, type 2 diabetes) before pregnancy
* Having a psychiatric diagnosis,
* Having a chronic disease
* Having risk factors such as threat of premature birth, placenta previa, premature rupture of membranes
* Having any disability that would prevent communication (deafness, hearing impairment, etc., use of languages other than Turkish),
* Pregnant women who do not want to continue the study and give birth before the 37th week of pregnancy will be excluded from the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2023-06-06 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-09-20 (Actual)

PRIMARY OUTCOMES:
Self-Efficacy Scale in Health Management | As the score obtained from the scale increases, self-efficacy for health practices increases.
  Before and after training between the 24th and 26th weeks of pregnancy
Quality of Life Scale | As the total score decreases, the quality of life decreases.
  Before and after training between the 24th and 26th weeks of pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Meltem Akbaş, PhD, Principal Investigator — Universty Of Cukurova
Locations (1):
- Meltem Akbaş, Adana, Sarıçam, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No